CLINICAL TRIAL: NCT04049357
Title: Colon Capsule Endoscopy in Bowel Cancer Screening. A Randomized Controlled Trial
Brief Title: Care for Colon 2015
Acronym: CFC2015
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 0
Record Dates: First submitted 2019-08-05; First posted 2019-08-08 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer; Adenoma
Keywords: Camera Capsule Endoscopy; Colorectal cancer screening; Optical colonoscopy; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Adenoma | interventions — Endoscopy

STUDY DESIGN:
Intervention Model Description: The investigators will include 124.214 consecutive citizens from the Region of Southern Denmark when they are invited for screening. The participants will be randomized into two groups using an automated randomization tool provided by Odense Patient data Explorative Network (OPEN). The randomization will be based on Zelen's pre-randomization principle and will take place prior to citizens receiving the invitation. The individuals are randomized into 62.107 people allocated in the intervention group and 62.107 allocated in the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- The intervention group (Experimental): If the FIT test is returned and positive the individual can choose either Camera Capsule Endoscopy (CCE) or Optical colonoscopy (OC) as the primary bowel investigation. If OC is chosen, it is performed as standard and the participant outcomes remains analyzed in the intervention group as intention to treat.
  If CCE is chosen an out-clinic CCE will be done at one of four regional sites. Overall and segmental bowel preparation grade (Leighton-Rex 1-4) and all pathological findings are reported. If the anal verge is identified without video blackout in the colon the transit is considered complete. Any incomplete CCE investigation will be followed by standard optical endoscopy to the extent needed to investigate the proportion of the colon not visualized by the capsule and remove any detected polyps. If the CCE is complete with complete transit and adequate preparation, individuals with more than two polyps or one polyp over 9 mm will be referred for colonoscopy.
  Interventions: Device: Camera Capsule Endoscopy/ PillCam
- The control group (No Intervention): The control group will be invited to screening as usual. The intervention group will be informed that if the fecal test is returned and positive they can either choose to have an initial colon capsule endoscopy, and only colonoscopy if significant findings are made or an initial colonoscopy as usual.

INTERVENTIONS:
Device: Camera Capsule Endoscopy/ PillCam — Camera Capsule Endoscopy in screening
  Arms: The intervention group

SUMMARY:
The investigatior believe that implementing camera capsule endoscopy as a filter test to colonoscopy will increase screening participation, increase the number of individuals with detected intermediate- high risk adenomas or cancer, reduce the colonoscopy demand and reduce the number of complications.

DETAILED DESCRIPTION:
The Danish national colorectal cancer screening program includes all citizens aged 50-74 years, who are invited biennially to a fecal test for invisible blood in the stool. If the test is positive the citizen is invited for a colonoscopy. 90% of the test-positive undergo colonoscopy. The detected cancers are at a significant earlier stage and survival from screening detected cancer is higher. It is also expected that cancer incidence will drop due to removal of the advanced adenomas before they develop into cancer. Although initial results are positive, there is room for improvement. Additionally there are rare but serious complications to colonoscopy in the form of bleeding or bowel perforation.

Through four years the investigators have tested the colon capsule endoscopy method, and find that the investigation is associated with significantly less discomfort and that the diagnostic ability to find polyps > 1 cm is better than colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Danish colorectal screening program

Exclusion Criteria:

* None

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2031 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
CCE detection rate of polyps compared to OC | Within 30 days
  The investigators aim to conduct a large scale randomized trial to investigate the implementation of CCE as part of the Danish screening protocol.

CONTACTS AND LOCATIONS:
Locations (1):
- Odense University Hospital, Svendborg Sygehus, Svendborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deding U, Boggild H, Baatrup G, Kaalby L, Hjelmborg J, Thygesen MK, Schelde-Olesen B, Kobaek-Larsen M; CareForColon2015 study group. Socioeconomic differences in expected discomfort from colonoscopy and colon capsule endoscopy. Prev Med. 2023 Aug;173:107593. doi: 10.1016/j.ypmed.2023.107593. Epub 2023 Jun 24. PMID 37364794
- [Background] Deding U, Boggild H, Kaalby L, Hjelmborg J, Kobaek-Larsen M, Thygesen MK, Schelde-Olesen B, Bjorsum-Meyer T, Baatrup G; CareForColon2015 study group. Socioeconomic differences in discrepancies between expected and experienced discomfort from colonoscopy and colon capsule endoscopy. Heliyon. 2024 Jul 8;10(14):e34274. doi: 10.1016/j.heliyon.2024.e34274. eCollection 2024 Jul 30. PMID 39100485
- [Background] Baatrup G, Bjorsum-Meyer T, Kaalby L, Schelde-Olesen B, Kobaek-Larsen M, Koulaouzidis A, Kroijer R, Al-Najami I, Buch N, Hogh A, Qvist N, Thygesen MK, Deding U; CareForColon2015 study group. Choice of colon capsule or colonoscopy versus default colonoscopy in FIT positive patients in the Danish screening programme: a parallel group randomised controlled trial. Gut. 2025 Sep 8;74(10):1616-1623. doi: 10.1136/gutjnl-2024-333687. PMID 40210462
- [Background] Deding U, Bjorsum-Meyer T, Kaalby L, Kobaek-Larsen M, Thygesen MK, Madsen JB, Kroijer R, Baatrup G. Colon capsule endoscopy in colorectal cancer screening: Interim analyses of randomized controlled trial CareForColon2015. Endosc Int Open. 2021 Nov 12;9(11):E1712-E1719. doi: 10.1055/a-1546-8727. eCollection 2021 Nov. PMID 34790535
- [Background] Kaalby L, Deding U, Kobaek-Larsen M, Havshoi AV, Zimmermann-Nielsen E, Thygesen MK, Kroeijer R, Bjorsum-Meyer T, Baatrup G. Colon capsule endoscopy in colorectal cancer screening: a randomised controlled trial. BMJ Open Gastroenterol. 2020 Jun;7(1):e000411. doi: 10.1136/bmjgast-2020-000411. PMID 32601101
- [Derived] Schelde-Olesen B, Koulaouzidis A, Deding U, Toth E, Dabos KJ, Eliakim A, Carretero C, Gonzalez-Suarez B, Dray X, de Lange T, Beaumont H, Rondonotti E, Kopylov U, Ellul P, Perez-Cuadrado-Robles E, Robertson A, Stenfors I, Bojorquez A, Piccirelli S, Raabe GG, Margalit-Yehuda R, Barba I, Scardino G, Ouazana S, Bjorsum-Meyer T. Bowel cleansing quality evaluation in colon capsule endoscopy: what is the reference standard? Therap Adv Gastroenterol. 2024 Oct 23;17:17562848241290256. doi: 10.1177/17562848241290256. eCollection 2024. PMID 39449979